CLINICAL TRIAL: NCT01308255
Title: A Multi-centre Randomised Double Blind Placebo Controlled Study Comparing Two Regimens of Combination Therapy in Early DMARD Naive Rheumatoid Arthritis.
Brief Title: Infliximab as Induction Therapy in Early Rheumatoid Arthritis (IDEA)
Acronym: IDEA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Paul Emery, Chief Investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RR05/7092; 2005-005013-37 (EudraCT Number)
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Methylprednisolone; Methylprednisolone Hemisuccinate; Methotrexate; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infliximab Arm (Experimental): For those randomised to the infliximab arm, infliximab will be administered at a dose of 3mg/kg according to the standard treatment protocol.
  Interventions: Drug: Infliximab; Drug: Methotrexate; Dietary Supplement: Folic acid
- Steroid/Placebo Arm (Placebo Comparator): Patients randomised to this arm will receive an IV infusion of 250mg methylprednisolone at week 0 & those without an adequate clinical response after 26 wks will receive additional steroid as IM methylprednisolone 120mg. Patients on this arm will receive an IV placebo infusion of 250ml of 9mg/l NaCl.
  Interventions: Drug: Methylprednisolone; Drug: Methotrexate; Dietary Supplement: Folic acid

INTERVENTIONS:
Drug: Infliximab — Prior to week 26
  * Infliximab 3mg/kg standard regime (weeks 0, 2, 6, 14, 22)
  * Methotrexate commencing at 10mg weekly, progressing to 20mg by week 6.
  * Folic acid 5 mg daily except the day methotrexate is taken
  Patients will be unblinded at week 26 and then treated pragmatically guided by disease activity
  Other Names: Remicade
  Arms: Infliximab Arm
Drug: Methylprednisolone — Steroid
  Other Names: Medrol, Solu-Medrol and Cadista.
  Arms: Steroid/Placebo Arm
Drug: Methotrexate — All patients enrolled are commenced on oral methotrexate 10mg once a week The methotrexate dose should be increased to 15 mg at the week 2 visit. The methotrexate should be increased to 20mg at the week 6 visit.
  Other Names: Maxtrex
Dietary Supplement: Folic acid — All patients enrolled are commenced on oral folic acid 5mg daily, except the day methotrexate is taken, and the study infusions.
  Other Names: vitamin B9,vitamin Bc, or folacin

SUMMARY:
This is a placebo controlled randomised clinical trial.Patients attending Yorkshire Early Arthritis Clinics and diagnosed with rheumatoid arthritis with symptom duration of 3-12 months will be recruited. They will be randomised to blinded therapy with either methotrexate and intravenous corticosteroid at baseline, or methotrexate and intravenous infliximab according to the standard treatment regime. Patients will be followed regularly, and at each visit, if the patients are not in remission, they will be given an intramuscular injection of corticosteroid. After 26 weeks, all patients will be unblinded and those with an inadequate treatment response will be treated according to a dose escalation algorithm until they achieve remission. Those in remission will continue on blinded therapy and if 6 months of remission is achieved the intravenous agent (infliximab or placebo) will be withdrawn.

DETAILED DESCRIPTION:
The main aim of the study is to compare the efficacy of biologic therapy (infliximab) as induction therapy against current best practice therapy: early introduction of methotrexate in combination with steroid induction therapy and dose modification according to predefined disease activity measures (as informed by the literature, and based around a pragmatic dose escalation protocol).

Exploratory analyses of imaging findings will be undertaken on a subgroup of patients at sites able to perform such assessments.

The imaging techniques used include

1. DEXA
2. US
3. Peripheral MRI

End point

The end points of the study are defined as:

* Completion of 78 weeks of therapy in the study
* Withdrawal due to any reason including toxicity or inefficacy
* Withdrawal due to completion of the dose escalation regime and disease remains active
* Withdrawal due to meeting NICE criteria for biologics during the dose escalation regime

At the end of the study, patients will continue to be followed in the Yorkshire Rheumatology clinics as part of their routine care.

All patients who withdraw will be asked to have a withdrawal visit with X-Rays of hands and feet to allow assessment of the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Men & Women 18-80 years of age.
* Fulfil 1987 ACR criteria for RA.
* Symptoms of > 3 months and < 12 months duration.
* Men and women must use adequate birth control measures for the duration of the study and should continue such precautions for 6 months after receiving the last infusion or dose of methotrexate.
* The patient must be able to adhere to the study visit schedule and other protocol requirements.
* The patient must be capable of giving informed consent and the consent must be obtained prior to any screening procedures.
* Must have a chest radiograph within 3 months prior to first treatment dose with no evidence of malignancy, infection or fibrosis.
* Are considered eligible according to the tuberculosis (TB) eligibility assessment.
* Active disease as defined by DAS > 2.4.
* TNF therapy naïve.
* DMARD therapy naïve.
* Negative hepatitis B and C screening tests within 3 months prior to screening.

Exclusion Criteria:

* Women who are pregnant, nursing, or men or women planning pregnancy within 24 months after screening.
* Use of any investigational (unlicensed) drug within 1 month prior to screening or within 5 half-lives of the investigational agent, whichever is longer.
* Previous or current treatment with any other therapeutic agent targeted at reducing TNF.
* Prior treatment with any DMARD.
* Serious infections (such as pneumonia or pyelonephritis) in the previous 3 months.
* Documented HIV infection.
* Hepatitis- B or Hepatitis-C serology positive (must be checked within 3 months prior to screening).
* Are considered ineligible according to the TB eligibility assessment.
* Have or have had an opportunistic infection within 6 months prior to screening.
* Significant haematological or biochemical abnormality.
* Have current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease.
* Concomitant congestive heart failure, including medically controlled asymptomatic patients.
* Presence of a transplanted organ (with the exception of a corneal transplant > 3 months prior to screening).
* Malignancy within the past 5 years.
* History of lymphoproliferative disease including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease.
* Known recent substance abuse (drug or alcohol).
* Poor tolerability of venipuncture or lack of adequate venous access for required blood sampling during the study period.
* Have a chest radiograph at screening that shows evidence of malignancy, infection, or any abnormalities suggestive of TB.
* Have a positive Mantoux test or evidence of active TB infection, or recent close contact with an individual with active TB.
* Previous oral, IM, IA or IV corticosteroids within 1 month prior to baseline.
* Receiving treatment with anakinra.
* Contra-indications to methotrexate, infliximab or steroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2006-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the change in Sharpe van der Heijde score | 50 Weeks

SECONDARY OUTCOMES:
Number of patients having a major clinical response (DAS <1.6 for 6 months) | 78 Weeks
The change in Sharpe van der Heijde scores between baseline, 26 & 72 wk hand & feet x-rays | Week 72
The number of patients in clinical remission (DAS <1.6) at 78 weeks | 78 Weeks
The number of patients in infliximab free remission (DAS <1.6) at 78 weeks | 78 Weeks
The number of patients in clinical remission (DAS <1.6) at 26 weeks | 26 Weeks
RA Quality of Life questionnaire | 78 Weeks
Health Assessment Questionnaire | 78 Weeks
Immunogenetic studies to predict long-term immune response | 78 Weeks
Immune phenotyping (flow cytometry) and assessment of immune effector & regulatory functions | 78 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul Emery, Principal Investigator — University of Leeds
Locations (1):
- Chapel Allerton Hospital, Leeds, West Yorkshire, United Kingdom